CLINICAL TRIAL: NCT04496596
Title: A Prospective, Double-Blind, Placebo-controlled Study of Suramin in Subjects With Furosemide-Resistant Acute Kidney Injury (AKI): Efficacy in Preventing Dialysis Dependent AKI
Brief Title: Study of Suramin in Subjects With Furosemide-Resistant AKI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rediscovery Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RLS003-02-001
Record Dates: First submitted 2020-07-29; First posted 2020-08-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Suramin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Suramin (Experimental)
  Interventions: Drug: Suramin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Suramin — Suramin is administered via IV infusion as a single dose of 3 mg/kg
  Arms: Suramin
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a prospective, double-blind, randomized, placebo-controlled study to assess the effects of suramin as a potential treatment option to prevent subjects with AKI from progressing to Kidney Disease Improving Global Outcomes (KDIGO) Stage III or dialysis dependent AKI.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age at the time of signing the informed consent
* KDIGO Stage I AKI and a serum Cr increase ≥ 0.3 mg/dL within 48 hr or 1.5 to 1.9-times baseline (pre-FST) Cr levels within 48 hr (± 6 hr) prior to randomization OR KDIGO Stage II AKI and serum Cr increase 2.0 to 2.9-times baseline (pre-FST) Cr levels within 48 hr (± 6 hr) prior to randomization
* Fails to achieve a 200 mL increase in urine output within 2 hr following a 1.0 mg/kg bolus of furosemide (i.e., positive FST)
* If female of childbearing potential, must have a negative pregnancy test at Screening Is capable of providing informed consent as described in in this protocol.

Exclusion Criteria:

* Receiving hemodialysis or peritoneal dialysis
* Prior renal transplant (other organ transplants are not excluded)
* Known baseline (pre-FST) estimated glomerular filtration rate (eGFR) ≤ 20 mL/min
* Evidence of hydronephrosis or obstructive uropathy confirmed by renal ultrasound (for subjects without a documented ultrasound, the
* Investigator will determine if a renal ultrasound is indicated, consistent with the standard of care (SOC)
* Hepatic encephalopathy, Child class C cirrhosis, and/or clinical suspicion of hepatorenal syndrome
* International normalized ratio (INR) ≤ 3.0, unless on stable long-term warfarin therapy within 2 weeks prior to randomization
* Known human immunodeficiency virus (HIV), hepatitis B or hepatitis C infection
* Known coronavirus (COVID-19) infection
* White blood cell count (WBC) < 2,000/μL and/or platelet count < 30,000/μL at the time of Screening
* A sequential organ failure assessment (SOFA) score > 10 during Screening
* Subjects requiring 3 or more vasopressor agents of any combination to maintain a mean arterial pressure > 65 mm Hg
* Unwilling to participate in follow-up phone surveys up to 180 days post-treatment
* Are enrolled in another interventional research study or have participated in another interventional study within 14 days of Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-12-22 (Estimated)

PRIMARY OUTCOMES:
To evaluate and compare the efficacy of a single 3.0 mg/kg infusion of suramin versus placebo in subjects with diuretic unresponsive AKI | 7 days
  The difference between the effect of a 3.0 mg/kg infusion of suramin versus placebo will be based on meeting 2 or more of the composite event endpoints of: peak serum creatinine (Cr) of 6 mg/dL or above from investigational product (IP) infusion through Day or progression to KDIGO Stage III within 72 hours (hr) from IP infusion or death or dialysis from IP infusion through Day 7.

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - University of Arkansas Medical Sciences (UAMS), Little Rock, Arkansas
  - California Institute of Renal Research, La Mesa, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Emory University School of Medicine, Atlanta, Georgia
  - Emory Johns Creek Hospital, Johns Creek, Georgia
  - University of Kentucky, Lexington, Kentucky
  - University of Missouri - Dept. of Surgery, Columbia, Missouri
  - University of New Mexico Health Science Center, Albuquerque, New Mexico
  - New York-Presbyterian Medical Center of Queens, Flushing, New York
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Southeast Renal Research Institute, Chattanooga, Tennessee
  - Baylor Scott and White Research Institute - Dallas Clinical Trials Office, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No